CLINICAL TRIAL: NCT00524381
Title: The Effect of Etanercept on the Early Clinical Course of Polymyalgia Rheumatica (Pilot Study)
Brief Title: Etanercept Treatment in the Early Course of Polymyalgia Rheumatica
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Professor Henrik Galbo, Department of Rheumatology, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMR-ENBREL-1
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Etanercept (Enbrel) — TNF-alpha antagonist, subcutaneous injection, 25 mg twice/week, 14 days.
Drug: Sodium chloride (placebo) — NaCl, isotonic saline, subcutaneous injection, 1 ml twice/week, 14 days.

SUMMARY:
The purpose of this study is to evaluate the effect of the tumor necrosis factor alpha (TNF) antagonist, etanercept, on the early clinical course of polymyalgia rheumatica (PMR).

PMR is a common inflammatory disease with an unknown etiology that is characterized by aching, tender, and stiff proximal muscle. Some evidence suggests that TNF plays a central role in the pathophysiology of PMR.

The preferred treatment with glucocorticoids (GCs) is adequate for most patients, but a subset of patients have a more prolonged, relapsing disease course. These patients require treatment with GCs for 1 to 2 years. GC related adverse events are frequent during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persons with active polymyalgia rheumatica (patients only).
* Signed informed consent and written authorization.

Exclusion Criteria:

* Other inflammatory conditions than polymyalgia rheumatica, including symptoms of giant cell arteritis, e.g. head aches, jaw claudication and visual disturbances.
* Current malignancy or history of malignancy.
* Neuromuscular conditions.
* Infections with systemic impact.
* Uncontrolled diabetes mellitus.
* Uncontrolled hypertension.
* Current tuberculosis or history of tuberculosis.
* Severe heart failure (NYHA class 3 and 4).
* Current use of glucocorticoids, biological drugs, and immunosuppressive drugs.

Exclusion Criteria (controls):

* Polymyalgia rheumatica.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Polymyalgia rheumatica activity score (PMR-AS) | 14 days

SECONDARY OUTCOMES:
Plasma concentrations of various cytokines, chemokines, and adipokines | 14 days
Quantitative use of analgesics | 14 days
Insulin sensitivity (HOMA) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Galbo, Professor, Study Director — Bispebjerg Hospital, Department of Rheumatology
Locations (1):
- Bispebjerg Hospital, Department of Rheumatology, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Kreiner FF, Galbo H. Activity of the neuroendocrine axes in patients with polymyalgia rheumatica before and after TNF-alpha blocking etanercept treatment. Arthritis Res Ther. 2012 Aug 15;14(4):R186. doi: 10.1186/ar4017. PMID 22894827
- [Derived] Kreiner F, Galbo H. Effect of etanercept in polymyalgia rheumatica: a randomized controlled trial. Arthritis Res Ther. 2010;12(5):R176. doi: 10.1186/ar3140. Epub 2010 Sep 20. PMID 20854662